CLINICAL TRIAL: NCT07150390
Title: Aetiologies and Prognosis of Small Bowel Obstruction in Virgin Abdomen
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiaochun Ping, Associate Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2023-SR-340
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Small Bowel Obstruction; Small Bowel Obstruction Adhesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBO-VA: small intestinal obstruction patients without a history of abdominal surgery (virgin abdomen)

SUMMARY:
Small bowel obstruction (SBO) is a surgical emergency in which the passage of intestinal contents is prevented due to mechanical obstruction of small intestine. It accounts for almost 50% of all emergency laparotomies with significant in-hospital morbidity and costs. SBO has known to occur in patients who had no prior abdominal surgery, referring to as a virgin abdomen (VA). Nowadays, non-operative management comprising of bowel decompression, water-soluble contrast agents, and fluid resuscitation have been found safe and efficacious in 70% of SBOs caused by adhesions (ASBO). However, based on the assumption that SBO in the virgin abdomen (SBO-VA) is usually caused by other aetiologies than adhesions, such as malignancy and hernias, many authors suggest that surgical exploration is still mandatory. Besides, recent studies do show high incidence of adhesions also in patients with SBO-VA. This observation signifies that guideline on the management of ASBO might also apply to the majority of patients with SBO-VA. Hence, the aim of our retrospectively study is to shed light on the aetiologies of SBO-VA. We believe treatment strategy needs to be based on the underlying reasons of obstructions and conditions of the patients and evaluate their prognosis accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Only patients without prior abdominal operations and with CT or surgical exploration confirmation of the diagnosis of SBO were included.

Exclusion Criteria:

* Patients with age less than 14 years were excluded in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2009 to December 2020, 2098 consecutive patients with 2275 admissions who diagnosed with bowel obstuction were enrolled in the First Affiliated Hospital of Nanjing Medical University, P. R. China. For patients with multiple admissions, only the index admissions were included, the rest were used for follow-up analysis. The detailed medical records of those 2098 patients were collected and reviewed. Only patients without prior abdominal operations and with CT or surgical exploration confirmation of the diagnosis of SBO were included. In addition, patients with age less than 14 years were excluded in this study. The diagnosis of SBO was established if an attending surgeon documented interpretation of CT imaging and was in agreement with the diagnosis. Finally, 312 patients with SBO in virgin abdomen were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The recurrence rate within 5 years after discharge | 5 years
  The recurrence rate of small bowel obstruction within 5 years after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided